CLINICAL TRIAL: NCT02993952
Title: Transcranial Direct Current Stimulation (tDCS) and Its Therapeutic Effects in Chikungunya Fever
Brief Title: tDCS and Its Therapeutic Effects in CK Fever
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio Grande do Norte (Other)
Responsible Party: Principal Investigator, Edson meneses da silva filho, Principal Investigator, Universidade Federal do Rio Grande do Norte
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1.839.742
Record Dates: First submitted 2016-12-05; First posted 2016-12-15 (Estimated); Last update posted 2017-04-18 (Actual); Status verified 2017-04

CONDITIONS: Chikungunya Fever
MeSH Terms: conditions — Chikungunya Fever | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active stimulation (Active Comparator): A constant current (anodic) of 2mA will be applied for 20 minutes on the Primary motor cortex.
  Interventions: Device: Transcranial Direct Current Stimulation
- Sham stimulation (Sham Comparator): A constant current (sham) of 2mA will be applied, but the stimulator will be turned off after 30 seconds on the Primary motor cortex.
  Interventions: Device: Sham Transcranial Direct Current Stimulation

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation — For electrode placement, the criteria used by the 10/20 electroencephalography system will be obeyed and the electrodes will be positioned area C3 for the anode and Fp2 (contralateral supraorbital area) for the cathode electrode. A constant current of 2mA will be applied for 20 minutes.
  Arms: Active stimulation
Device: Sham Transcranial Direct Current Stimulation — For electrode placement, the criteria used by the 10/20 electroencephalography system will be obeyed and the electrodes will be positioned area C3 for the anode and Fp2 (contralateral supraorbital area) for the cathode electrode, but the stimulator was turned off after 30 seconds of stimulation. Therefore, patients in the sham group felt the initial itching sensation but received no current for the rest of the stimulation period.
  Arms: Sham stimulation

SUMMARY:
One of the major challenges faced by researchers working in the field of rehabilitation science is the ability to provide integrative approaches to the use of clinical practice. In this context it becomes increasingly necessary to construct investigative approaches, so that they can reach clinical practice in a shorter period of time,since the large volume of information produced globally does not impact in the short or medium term on new therapeutic recommendations. Among the various chronic painful entities, there is chikungunya fever as a highlight for having a rich clinical chronology in relation to pain. Its therapy is used done by drugs in almost all national and international consensuses, therefore therapy against pain in chikungunya fever is limited during the rehabilitation process. It is very important that the science of rehabilitation enhances methods of noninvasive brain modulation that enable, through the excitation or inhibition of specific cortical areas to produce pain inhibiting effects, providing a simple and low cost treatment to the clinical routine.Technological advances and non-invasive techniques to modulate brain function have been developed, for instance, Transcranial Direct Current Stimulation (tDCS).

The objective of the present project is to present the tDCS as a new modality of physical rehabilitation for the patient with chronic pain resulting from chikungunya fever. The purpose of the study is to present physical, behavioral and social results of the application of tDCS in chikungunya fever, suggesting an improvement in the quality of life and functional status of the individual.

ELIGIBILITY:
Inclusion Criteria:

* Laboratory or medical diagnosis of chikungunya fever, being in the chronic phase of the disease, intellectual and physical capacity preserved for conducting research tests.

Exclusion Criteria:

* History of seizures or epileptic disease, pregnancy, states associated with other previously diagnosed rheumatic diseases such as rheumatoid arthritis, gout and lupus, under 18 years and over 65 of age, patients with signs of severity and/or indication for hospitalization.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-12-12 (Actual); Primary Completion 2017-02-20 (Actual); Study Completion 2017-03-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline Pain at 3 weeks | Every day during 3 weeks (before treatment, during treatment and one week after treatment).
  Diary of pain
Change from baseline Pain at 3 weeks | baseline (one week before starting stimulation), one week after baseline (after first stimulation), eleven days after baseline (after last stimulation) and 3 weeks after baseline.
  Visual analogue scale.
Change from baseline Pain at 3 weeks | baseline (one week before starting stimulation), one week after baseline (after first stimulation), eleven days after baseline (after last stimulation) and 3 weeks after baseline.
  Diagnosing Neuropathic Pain - DN4 Questionnaire
Change from baseline Pain at 3 weeks | baseline (one week before starting stimulation), one week after baseline (after first stimulation), eleven days after baseline (after last stimulation) and 3 weeks after baseline.
  McGill Pain Questionnaire short brazilian version (Br- MPQ)
Change from baseline Pain at 3 weeks | baseline (one week before starting stimulation), one week after baseline (after first stimulation), eleven days after baseline (after last stimulation) and 3 weeks after baseline.
  Brief Pain Inventory (Short Form).

SECONDARY OUTCOMES:
Change from baseline Quality of Life at 3 weeks | baseline (one week before starting stimulation), one week after baseline (after first stimulation), eleven days after baseline (after last stimulation) and 3 weeks after baseline.
  Short Form 36 Health Survey (SF-36).
Change from baseline Flexibility at 3 weeks | baseline (one week before starting stimulation), one week after baseline (after first stimulation), eleven days after baseline (after last stimulation) and 3 weeks after baseline.
  Sit and Reach Flexibility Test.
Change from baseline Flexibility at 3 weeks | baseline (one week before starting stimulation), one week after baseline (after first stimulation), eleven days after baseline (after last stimulation) and 3 weeks after baseline.
  Back Scratch Test.
Change from baseline Strength at 3 weeks | baseline (one week before starting stimulation), one week after baseline (after first stimulation), eleven days after baseline (after last stimulation) and 3 weeks after baseline.
  The 30-Second Chair Stand Test.
Change from baseline Strength at 3 weeks | baseline (one week before starting stimulation), one week after baseline (after first stimulation), eleven days after baseline (after last stimulation) and 3 weeks after baseline.
  Elbow flexion strength test
Change from baseline Strength at 3 weeks | baseline (one week before starting stimulation), one week after baseline (after first stimulation), eleven days after baseline (after last stimulation) and 3 weeks after baseline.
  Manual Muscle Testing (Hand Dynamometer)

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo Pegado Freitas, PhD, Study Director — Universidade Federal do Rio Grande do Norte; Edson Meneses Filho, Graduate, Principal Investigator — Universidade Federal do Rio Grande do Norte
Locations (1):
- Federal University of Rio Grande do Norte, Santa Cruz, Rio Grande do Norte, Brazil

IPD SHARING:
Plan to Share IPD: No